CLINICAL TRIAL: NCT03947892
Title: Predictive Value of PET CT in the Histologic Lymph Node Status of Patients With Squamous Cell Carcinoma of the Oral N0 Clinical and Radiological Cavity.
Acronym: ORNICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.064; 2019-A00883-54 (Other: ID RCB)
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Squamous Cell Carcinoma of the Oral; Clinically Node-Negative and Radiology
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET-CT — A PET-CT scan will be performed systematically for all patients included with the SUVmax, SUV peak, MTV of the lesion, and up to 3 suspicious ganglia during the visual analysis.

SUMMARY:
Squamous cell carcinoma of the VADS represents the majority of cancers in ENT. Metastatic lymph node involvement is an important prognostic factor. In N0 patients clinically and scanographically, the prevalence of cervical lymph node metastasis remains important. Only the anatomopathological analysis of cervical lymph node dissection confirms the presence of a micro-metastasis. However, new criteria of interpretation in nuclear medicine seem promising in the detection of lymph node lesions not detectable in traditional imaging.

The main objective of this study is to study the positive predictive value (PPV) of CT scans in the anatomo-pathological analysis of N0 clinical and radiological or N + unilateral neck ganglia in patients with squamous cell carcinoma of the oral cavity.

DETAILED DESCRIPTION:
The main objective is to study the positive predictive value of PET-CT in the identification of infra-clinical lymph node lesions for cancers of the oral cavity classified N0 or N + unilateral

Patients are admitted to ORL or maxillofacial consultation with initial clinical examination according to current recommendations (tumor evaluation, cervical palpation, locoregional examination).

A dated and signed diagram of the lesion and ganglionic areas will be made during this consultation.

A biopsy for histopathological examination of the lesion will be necessary to confirm the diagnosis of squamous cell carcinoma with P16 analysis. It will be performed during the consultation under local anesthesia if the lesion is accessible or under general anesthesia during panendoscopy.

All patients will benefit from an assessment of locoregional extension by CT cervicofacial and thoracic injected (in order to look for possible pulmonary metastases or suspicious mediastinal lymphadenopathies) as requested in the oncological recommendations and PET-CT. As part of the extension assessment, a panendoscopy or bronchial fibroscopy and gastro-oesophageal failure will be performed if risk factors ethanolotagagic are present.

If the lesion is not accessible for a biopsy during the inclusion visit, the patient is summoned for a panendoscopy. It is an examination under general anesthesia to make a biopsy of the primary tumor and to search for the absence of synchronous localization. In current practice, this examination requires overnight hospitalization.

The patient will be reviewed by the ORL or maxillofacial surgeon in consultation after receiving the anatomopathological findings of the lesion and the entire extension assessment (CT cervico-thoracic injected and PET-CT).

On CT PET, an analysis with additional interpretation criteria will be performed (SUVmax, SUV peak, MTG) on the primary tumor and on the invaded lymph nodes. A ganglion is considered invaded when its SUV is suppressed at 30% of the SUV of the original lesion.

The patient's file will have been previously presented in a Multidisciplinary Concertation Meeting, whose treatment will consist of a surgical excision of the primary lesion and a lymph node dissection.

The patient will be seen again in consultation at 10 days of his intervention as part of the follow-up postoperative in order to be able to receive all the anatomopathologic results of the operative specimen and ganglion dissection. The patient's record will have been represented in CPR in order to decide whether or not to have an adjuvant treatment based on the anatomopathological characters (capsular rupture, number of ganglions invaded, peri-nervous sheath).

ELIGIBILITY:
Inclusion Criteria:

* 1st localization of squamous cell carcinoma of the oral cavity.
* Any tumor T according to the 2017 classification, N0 clinical and radiological or N + unilateral, M0
* Not challenged for tumor resection surgery and bilateral dissection.

Exclusion Criteria:

* age <18 years
* opposition of the curator concerning the person under guardianship
* subject under guardianship or deprived of liberty
* antecedent treatment of cancer of the upper aero-digestive tract (surgery, radiotherapy, chemotherapy)
* any current treatment for another cancer site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population selected is that of any patient with squamous cell carcinoma of the oral cavity classified N0 clinical and radiological or unilateral N +, M0, not challenged for tumor resection surgery and bilateral cervical dissection. They will benefit in their assessment of extension of a PET-CT.
  Patients will be selected during an ENT or maxillofacial consultation. They will receive clear and appropriate information from the study. They will decide whether to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
metastatic lymph node involvement | 30 days
  The outcome is analyzing histologic metastatic lymph node. The outcome data table will include the presence of histologic metastatic lymph node, localization of the lymph invaded, presence of capsular rupture, and preoperative TEP CT data.

CONTACTS AND LOCATIONS:
Overall Officials: Claire DUCROZ, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Arya S, Rane P, Deshmukh A. Oral cavity squamous cell carcinoma: role of pretreatment imaging and its influence on management. Clin Radiol. 2014 Sep;69(9):916-30. doi: 10.1016/j.crad.2014.04.013. Epub 2014 Jun 5. PMID 24908285
- [Background] Schoder H, Carlson DL, Kraus DH, Stambuk HE, Gonen M, Erdi YE, Yeung HW, Huvos AG, Shah JP, Larson SM, Wong RJ. 18F-FDG PET/CT for detecting nodal metastases in patients with oral cancer staged N0 by clinical examination and CT/MRI. J Nucl Med. 2006 May;47(5):755-62. PMID 16644744
- [Background] Ng SH, Yen TC, Chang JT, Chan SC, Ko SF, Wang HM, Lee LY, Kang CJ, Wong AM, Liao CT. Prospective study of [18F]fluorodeoxyglucose positron emission tomography and computed tomography and magnetic resonance imaging in oral cavity squamous cell carcinoma with palpably negative neck. J Clin Oncol. 2006 Sep 20;24(27):4371-6. doi: 10.1200/JCO.2006.05.7349. PMID 16983105
- [Background] Stoeckli SJ, Steinert H, Pfaltz M, Schmid S. Is there a role for positron emission tomography with 18F-fluorodeoxyglucose in the initial staging of nodal negative oral and oropharyngeal squamous cell carcinoma. Head Neck. 2002 Apr;24(4):345-9. doi: 10.1002/hed.10057. PMID 11933176
- [Background] Lee SJ, Choi JY, Lee HJ, Baek CH, Son YI, Hyun SH, Moon SH, Kim BT. Prognostic value of volume-based (18)F-fluorodeoxyglucose PET/CT parameters in patients with clinically node-negative oral tongue squamous cell carcinoma. Korean J Radiol. 2012 Nov-Dec;13(6):752-9. doi: 10.3348/kjr.2012.13.6.752. Epub 2012 Oct 12. PMID 23118574
- [Background] Ryu IS, Kim JS, Roh JL, Cho KJ, Choi SH, Nam SY, Kim SY. Prognostic significance of preoperative metabolic tumour volume and total lesion glycolysis measured by (18)F-FDG PET/CT in squamous cell carcinoma of the oral cavity. Eur J Nucl Med Mol Imaging. 2014 Mar;41(3):452-61. doi: 10.1007/s00259-013-2571-z. Epub 2013 Oct 1. PMID 24081448
- [Background] Chung MK, Jeong HS, Son YI, So YK, Park GY, Choi JY, Hyun SH, Kim HJ, Ko YH, Baek CH. Metabolic tumor volumes by [18F]-fluorodeoxyglucose PET/CT correlate with occult metastasis in oral squamous cell carcinoma of the tongue. Ann Surg Oncol. 2009 Nov;16(11):3111-7. doi: 10.1245/s10434-009-0621-3. Epub 2009 Jul 16. PMID 19609618